CLINICAL TRIAL: NCT01022060
Title: Efficacy of Renalof in the Dissolution of Renal Calculi in Patients With Recurrent Calcic Lithiasis
Brief Title: Renalof in the Dissolution of Renal Calculi in Patients With Recurrent Calcic Lithiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Mirna Atiés Sánchez, Institute of Nephrology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0913-CU
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Recurrent Calcic Urolithiasis
Keywords: Dietary supplement; Renalof; Recurrent calcic urolithiasis; Renal calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Renalof
  Interventions: Dietary Supplement: Renalof
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Renalof — One Renalof tablet (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 12 weeks
  Arms: A
Dietary Supplement: Placebo — One Placebo tablet (Orally administered) three time a day (just before each meal: breakfast, lunch and dinner), for 12 weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine whether Renalof administration promotes partial or total dissolution of urinary calculi and improves physicochemical parameters and metabolic activity in patients with recurrent calcic urolithiasis. The duration of this double-blind placebo controlled phase 3 clinical trial will be 12 weeks. The estimated number of patients to be recruited and randomized for the study is 110. Ultrasonographic and humoral parameters will be assessed every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic calcic lithiasis
* Calculus size lesser than or equal to 2.0 cm (0.79 inches)
* Signed informed consent

Exclusion Criteria:

* Calculus size greater than 2,0 cm (0.79 inches)
* Pregnancy
* Malignant neoplastic conditions
* Previous treatment for destruction of calculi in the urinary tract

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Size of calculi at week 12 (end of the treatment); week 0 refers to the beginning of treatment) | 12 weeks
Number of calculi at week 12 (end of the treatment); week 0 refers to the beginning of treatment | 12 weeks
Lithiasic activity at week 12 (end of the treatment); week 0 refers to the beginning of treatment | 12 weeks

SECONDARY OUTCOMES:
Calciuria at week 12 | 12 weeks
Uricosuria at week 12 | 12 weeks
Blood Uric acid at week 12 | 12 weeks
Oxaluria at week 12 | 12 weeks
Citraturia at week 12 | 12 weeks
Phosphatemia at week 12 | 12 weeks
Calcemia at week 12 | 12 weeks
Total plasmatic calcium at week 12 | 12 weeks
Blood ionic calcium at week 12 | 12 weeks
Calcium Oxalate crystallization risk at week 12 | 12 weeks
Calcium phosphate activity product at week 12 | 12 weeks
Calcium Oxalate activity product at week 12 | 12 weeks
pH of urine at week 12 | 12 weeks
Presence of adverse effects at any moment of treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mirna Atiés Sánchez, MD, Principal Investigator — Institute of Nephrology
Locations (1):
- Institute of Nephrology, Havana, La Habana, Cuba